CLINICAL TRIAL: NCT03506347
Title: Regional Prophylactic Vancomycin With Restricted Tourniquet Time in Primary Total Knee Replacement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark J. Spangehl, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-007853
Record Dates: First submitted 2018-04-17; First posted 2018-04-24 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Arthropathy of Knee Joint
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vancomycin 15mg/kg IV (Active Comparator): Will receive 15mg/kg based on actual body weight (maximum of 2g) of vancomycin via the systemic route at a rate of 15mg/kg as per hospital guidelines. Systemic IV vancomycin is given via a forearm vein, given over an infusion timed to finish immediately prior to surgery.
  Interventions: Drug: Vancomycin
- Vancomycin 500mg Intraosseous (Experimental): Will have the limb exsanguinated and an above knee tourniquet inflated to 300 mmHg. Immediately following tourniquet inflation, Group B will receive 500mg of vancomycin, via an EZ-IO intraosseous cannula. The vancomycin would be administered in 150ml of saline solution. The intraosseous cannula would be placed into the epiphysis of the proximal tibia. The tourniquet will be left inflated for 10 minutes following completion of the IORA injection then deflated.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Antibiotic
  Other Names: Vancocin

SUMMARY:
The purpose of this study is to determine whether or not giving a lower dose of antibiotics (Vancomycin) in the area where it is needed (the knee joint) is more effective at obtaining adequate tissue levels of the antibiotic than the current standard dose which is given intravenously (IV) through a wrist vein. The use of intraosseous regional administration (IORA) of vancomycin requires the use of a tourniquet for the duration of the procedure. Many surgeons prefer to perform the surgery with tourniquet use minimised or without a tourniquet at all. The aim of this study is to evaluate whether IORA vancomycin can achieve effective tissue concentrations with tourniquet use minimised.

DETAILED DESCRIPTION:
Patients are assigned to one of two groups by chance (like a coin toss):

GROUP A - Will receive 15mg/kg based on actual body weight (maximum of 2g) of vancomycin via the systemic route at a rate of 15mg/kg as per hospital guidelines. Systemic IV vancomycin is given via a forearm vein, given over an infusion timed to finish immediately prior to surgery.

GROUP B - Will have the limb exsanguinated and an above knee tourniquet inflated to 300 mmHg. Immediately following tourniquet inflation, Group B will receive 500mg of vancomycin, via an EZ-IO intraosseous cannula. The vancomycin would be administered in 150ml of saline solution. The intraosseous cannula would be placed into the epiphysis of the proximal tibia. The tourniquet will be left inflated for 10 minutes following completion of the IORA injection then deflated.

Both Groups will receive weight-based dose of systemic cefazolin ( or alternative antibiotic if allergic to cefazolin 15 minutes prior to inflation of tourniquet. This ensures all patients in the study receive effective antibiotic prophylaxis regardless of randomization. Both groups of patients would then undergo routine prep and draping For both groups, Total knee replacement would then be carried out as normal and the tourniquet will be inflated for cementation of the implants.

TISSUE SAMPLES Ten (10) tissue samples will be taken from each patient, 6 'fat' samples and 4 'bone' samples. Each sample is very small, around the size of a pinhead. Bone samples will be taken from the femur only to ensure no direct contamination from the site of injection (tibia) In addition, drain samples will be taken from the intra-articular drain site to measure vancomycin concentration the morning following surgery.

Three blood samples will be taken in both groups, intraoperatively, in recovery, and the following morning.

These samples are frozen and sent to a lab for analysis.

ELIGIBILITY:
Inclusion Criteria

Primary Total Knee Arthroplasty for osteoarthritis Informed consent given

Exclusion Criteria

Current or treatment with IV Vancomycin within preceding 7 days Previous hypersensitivity to vancomycin Significant cardiac or respiratory abnormality Patient has contraindications to IO vascular access using the EZ-IO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Spangehl, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spangehl MJ, Clarke HD, Moore GA, Zhang M, Probst NE, Young SW. Higher Tissue Concentrations of Vancomycin Achieved With Low-Dose Intraosseous Injection Versus Intravenous Despite Limited Tourniquet Duration in Primary Total Knee Arthroplasty: A Randomized Trial. J Arthroplasty. 2022 May;37(5):857-863. doi: 10.1016/j.arth.2022.01.057. Epub 2022 Jan 26. PMID 35091036
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin 500mg Intraosseous: Will have the limb exsanguinated and an above knee tourniquet inflated to 300 mmHg. Immediately following tourniquet inflation, Group B will receive 500mg of vancomycin, via an EZ-IO intraosseous cannula. The vancomycin would be administered in 150ml of saline solution. The intraosseous cannula would be placed into the epiphysis of the proximal tibia. The tourniquet will be left inflated for 10 minutes following completion of the intraosseous regional administration (IORA) injection then deflated.
  Vancomycin: Antibiotic
Period: Overall Study
Arm/Group | Vancomycin 15mg/kg IV | Vancomycin 500mg Intraosseous
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin 15mg/kg IV | Vancomycin 500mg Intraosseous | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8.29) | 69.1 (8.15) | 68 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Vancomycin Concentration in Fat
Description: Mean vancomycin concentration in fat measured in ug/g at surgical closure
Time Frame: Approximately 60 minutes post surgical incision
Measure: Mean (Standard Deviation); unit: ug/g
Units Other Than Participants: fat
Arm/Group | Vancomycin 15mg/kg IV | Vancomycin 500mg Intraosseous
Number analyzed (Participants) | 12 | 12
Number analyzed (fat) | 72 | 72
ug/g | 6.0 (0.85) | 40.5 (8.08)
Statistical Analysis 1: Comparison: Vancomycin 15mg/kg IV vs Vancomycin 500mg Intraosseous; Test type: Superiority; p = 0.001, ANOVA

2. Primary Outcome: Vancomycin Concentration in Bone
Description: Mean vancomycin concentration in bone measured in ug/g at surgical closure
Time Frame: Approximately 60 minutes post surgical incision
Measure: Mean (Standard Deviation); unit: ug/g
Units Other Than Participants: bone
Arm/Group | Vancomycin 15mg/kg IV | Vancomycin 500mg Intraosseous
Number analyzed (Participants) | 12 | 12
Number analyzed (bone) | 48 | 48
ug/g | 8.3 (0.77) | 26.9 (1.31)
Statistical Analysis 1: Comparison: Vancomycin 15mg/kg IV vs Vancomycin 500mg Intraosseous; Test type: Superiority; p = 0.009, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected from approximately 90 minutes prior to surgery to the morning after surgery for each subject, over the duration of approximately four months.
Arm/Group | Vancomycin 15mg/kg IV | Vancomycin 500mg Intraosseous
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03506347/Prot_SAP_000.pdf